CLINICAL TRIAL: NCT05741645
Title: The Effect of Elastic Banding on the Elasticity of the Lumbar Stabilizer Muscles in Individuals With Non-specific Low Back Pain.
Brief Title: Effect of Elastic Taping on Stiffness of Lumbar Stabilizer Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Lecturer, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-KAEK-120
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Study group consists of 15 participants, where the elastic kinesiotaping is applied and evaluations are made before and after.
  Interventions: Other: Kinesiotaping
- Control Group (Sham Comparator): To the participants in the control group, the elastic taping will be randomly applied to a place outside the area to be measured, without stretching, and without causing any effect.
  Interventions: Other: Sham Kinesiotaping

INTERVENTIONS:
Other: Kinesiotaping — During the kinesio taping of the erector spina vs multifidus muscles, the patient is in a standing position. Kinesiotape is applied with 50% tension and stays in the patient for 30 minutes.
  Arms: Study group
Other: Sham Kinesiotaping — The elastic taping will be randomly applied to a place outside the area to be measured, without stretching, and without causing any effect.
  Arms: Control Group

SUMMARY:
Low back pain is a common health problem worldwide. Epidemiological studies have shown that 70-80% of all people are affected at least once in their lifetime.

Although it is common, often the cause of the pain has not been determined and is called 'nonspecific low back pain. Chronic low back pain ranks second among the most common pain complaints under the age of 45 in the industrial age of limited activity. Organic pathology is not encountered in most musculoskeletal system pains. There are usually many underlying causes. The current literature offers a variety of treatment options, depending on the duration and severity of the symptoms of non-specific low back pain. These treatments include behavioral cognitive therapy, medication, electrophysical agents, manual therapy, and general exercises. Looking at the literature, it has been observed that there are not many objective studies investigating the effect of elastic bandage application on muscle elasticity.

'Shear Wave Elastography' is a method that quantitatively reveals the elasticity of tissues by measuring the speed of shear waves formed in the tissues through non-invasive high-frequency ultrasound waves. In recent studies, Shear Wave Elastography has shown promising results in demonstrating the elasticity of peripheral nerves.

ELIGIBILITY:
Inclusion Criteria:

* patients who diagnosed with non-specific low back pain
* between the ages of 18-24
* patients who able to perform at least 40° of trunk flexion

Exclusion Criteria:

* patients who obese, pregnant, had specific low back pain
* indication for surgery in the past 1 year
* the trauma of lumbar region, and systemic inflammatory disease affecting this area
* exercise and conventional physiotherapy in the last 6 months

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
muscle stiffness | 4 weeks
  The muscle stiffness of lumbar back muscles will be assessed using the B-mode of the ultrasound Shear Wave Elastography (SWE) imaging device. Longitudinal ultrasound Shear Wave Elastography images of the multifidus and erector spinal muscles will be taken bilaterally with a linear array probe in the prone position.

SECONDARY OUTCOMES:
The sit and reach test | 4 weeks
  The test is administered using the sit-and-reach test box. Subjects are seated on flat ground. The soles of both feet are flat on the test bench and the knees are asked to maintain contact with the ground in full extension. Participants are asked to reach forward on the measurement line with their palms facing down and hands on top of each other, and wait for a second or two at the last point they can reach with their hands; After three attempts, the best score is recorded. Foot level is considered 0, measurements that do not reach foot level are recorded as negative and values exceeding foot level are recorded as positive.
The functional reach test | 4 weeks
  It is applied to measure the functional balance of the individual and the amount of dynamic reach. Individuals are asked to reach as far as they can without their heels off the ground and without hip flexion.
Lateral bridge test | 4 weeks
  The participant lying on his/her non-dominant side will be asked to form a support surface from the elbow with the arm below, to place the other hand on the waist, and to build a bridge by raising the hip and knee. The time the balance is maintained will be recorded
The Flamingo Test | 4 weeks
  According to this test, the research group; 50 cm. in length, 4 cm. in height and 3 cm. Patient stands in balance by stepping on a wooden balance beam with his dominant foot. Bend the other foot at the knee and pull it towards the hip, holding it with the hand on the same side. While the research group is in balance with one leg in this way, the time starts and they try to stay balanced in this way for 1 minute. When the balance is disturbed (if he leaves while holding his foot, falls from the board, touches the ground with any part of his body, etc.), the time-time is stopped. When the research group regains its balance by climbing on the balance beam, the time continues from where it left off. The test continues in this way for one minute. When the time is up, each attempt to balance (after falling) by the research group is counted, and this number is recorded as the research group's score when the one minute time is up at the end of the test.
Back isometric endurance test | 4 weeks
  For this test, the participant is placed in a prone position with the torso hanging from the bed from the anterior superior iliac spine. The athlete is asked to keep his body parallel to the ground against gravity, with the legs fixed at the level of the gastrocnemius muscle and the hands clasped on the chest. Partial trunk extension is allowed. When the posture is disturbed and/or the athlete quits the experiment due to fatigue and pain, the time is stopped and the score in seconds is recorded.
Oswestry Disability Index | 4 weeks
  It consists of a total of 10 items measuring the severity of pain, personal care, lifting, walking, sitting, standing, social life, sleeping, traveling and the degree of pain. Each item is graded between 0-5. As the total score increases, the level of disability increases. The maximum score is 50 points; It is evaluated as heavy between 31-50 points, moderate between 11-30 points and mild between 1-10 points. The percentage of disability can be calculated by converting the total score obtained from the patient to the percentage system.
Visual Analogue Scale | 4 weeks
  Pain will be measured with a Visual Analogue Scale (VAS). VAS is the most commonly used method for measuring pain level. The score range is from 0 to 10. 0 points indicates no pain, 10 points unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No